CLINICAL TRIAL: NCT05928845
Title: Could Changes in Sternocleidomastoid Muscle Thickness be a Predictor of Sarcopenia in Intensive Care Patients?
Brief Title: Sternocleidomastoid Thickness in Sarcopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Asst. Prof., Namik Kemal University
Other Study IDs: 2022.67.04.17
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia
Keywords: sarcopenia; intensive care; ultrasonography
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Muscle thickness measurement: Rectus femoris and sternocleidomastoideus muscle thickness will be measured via ultrasonography
  Interventions: Diagnostic Test: Muscle thickness measurement

INTERVENTIONS:
Diagnostic Test: Muscle thickness measurement — Rectus femoris and sternocleidomastoideus muscle thickness will be measured via ultrasonography in admission and on 7th day of admission

SUMMARY:
In order to prevent sarcopenia in intensive care patients and to guide nutritional therapy, evaluation of muscle thickness with ultrasonography is a modern, simple and non-invasive procedure routinely performed by Anesthesiology and Reanimation specialists. Sarcopenia in intensive care patients has been demonstrated in many studies. It has been studied that routine examination of changes in rectus femoris muscle thickness by ultrasonography is a predictor of sarcopenia. However, the muscles in the neck region, such as the sternocleidomastoid muscle, which are easy to examine, have not been studied very well. There is no study in the literature with the sternocleidomastoid muscle. For this reason, we decided to examine the relationship of sternocleidomastoid muscle thickness with patient characteristics, treatments, feeding route and type, feeding time, length of stay in intensive care unit, as in routine measurements of rectus femoris muscle thickness by ultrasonography.

DETAILED DESCRIPTION:
Sarcopenia is an important clinical condition, characterized by a decrease in muscle mass and function that increases with age, especially in elderly patients. Studies have shown that sarcopenic patients have higher morbidity and mortality rates than non-sarcopenic patients. Along with the increased risk of muscle wasting in intensive care patients, there is an increase in both hospital mortality rates and the frequency of post-hospital mobilization problems.

Intensive care patients are a group of patients who are very prone to protein-energy malnutrition, and this leads to complications such as nosocomial infection and multiple organ failure, leading to prolongation of the stay in the intensive care unit, as well as an increase in morbidity and mortality. Therefore, nutritional support is a routine requirement of intensive care treatment and has a vital role in the prevention and treatment of nutritional deficiencies in intensive care patients.

The first point that should be evaluated in terms of the follow-up of a patient on whom nutritional support is maintained is to know for what reason, when, and what kind of treatment is planned in terms of quality and quantity. This is a starting point for monitoring. Knowing the patient's clinical and laboratory values when nutritional therapy is initiated allows the evaluation of how these data have changed during follow-up. The purpose of assessment of nutritional status is to identify the type and degree of malnutrition in order to make a rational treatment approach. However, there is no test that is both sensitive and specific to determine malnutrition in intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are expected to be followed up in the intensive care unit for at least 1 week
* Patients over 18 years old

Exclusion Criteria:

* Patients under 18 years of age
* Head-neck, femur trauma patients
* Those with a diagnosis of primary neuromuscular disease
* Those who have a condition that prevents imaging in the body parts where ultrasonography is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are expected to be followed up in the intensive care unit for at least 1 week in a tertiary university research and education hospital based 11 bed ICU
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | 1 week
  Rectus femoris and Sternocleidomastoideus muscle thickness change when compared to the value measured at admission to the intensive care unit.

SECONDARY OUTCOMES:
Nutrition regime | 1week
  Nutrition regimes, calorie and protein intake during admission will be saved.
Nutrition Scores | Day 1
  NRS 2002, NUTRIC scores will be calculated in admission

CONTACTS AND LOCATIONS:
Overall Officials: Onur Baran, Asst. Prof., Study Director — Department of Anesthesiology and Reanimation, Tekirdağ Namık Kemal University, Tekirdağ, Turkey; Ayhan Şahin, Asst. Prof., Principal Investigator — Department of Anesthesiology and Reanimation, Tekirdağ Namık Kemal University, Tekirdağ, Turkey; Cavidan Arar, Prof., Study Chair — Department of Anesthesiology and Reanimation, Tekirdağ Namık Kemal University, Tekirdağ, Turkey
Locations (1):
- Tekirdag Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kizilarslanoglu MC, Kuyumcu ME, Yesil Y, Halil M. Sarcopenia in critically ill patients. J Anesth. 2016 Oct;30(5):884-90. doi: 10.1007/s00540-016-2211-4. Epub 2016 Jul 4. PMID 27376823
- [Background] Rustani K, Kundisova L, Capecchi PL, Nante N, Bicchi M. Ultrasound measurement of rectus femoris muscle thickness as a quick screening test for sarcopenia assessment. Arch Gerontol Geriatr. 2019 Jul-Aug;83:151-154. doi: 10.1016/j.archger.2019.03.021. Epub 2019 Mar 27. PMID 31029040
- See also: Reference — https://pubmed.ncbi.nlm.nih.gov/27376823/